CLINICAL TRIAL: NCT03165786
Title: A Cognitive Behavioral Intervention to Reduce Fear of Hypoglycemia in Young Adults With Type 1 Diabetes
Acronym: FREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Pamela Martyn-Nemeth, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-0206
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Type1diabetes
Keywords: fear of hypoglycemia; self-management; glycemic control; glycemic variability

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FREE Group (Experimental): Cognitive behavioral therapy intervention with real-time continuous glucose monitoring.
  Interventions: Behavioral: FREE
- Control Group (No Intervention): Real-time continuous glucose monitoring

INTERVENTIONS:
Behavioral: FREE — Cognitive behavioral therapy with real-time continuous glucose monitoring.
  Other Names: CBT
  Arms: FREE Group

SUMMARY:
This study is being conducted to determine the feasibility of a cognitive behavioral therapy intervention to reduce fear of hypoglycemia and improve glucose levels in young adults with type 1 diabetes.

DETAILED DESCRIPTION:
In persons with type 1 diabetes (T1DM), iatrogenic hypoglycemia is the major limiting factor in achieving optimal blood glucose control. All persons with T1DM are at risk for hypoglycemia (blood glucose level < 70 mg/dl), which is life-threatening and has serious physical symptoms and psychological sequelae that lead to profound fear of future hypoglycemic events. This fear results in greater glucose variability (the intra-day fluctuations in blood glucose), due to under- or overcompensation of food intake, insulin dosing, or physical activity, as well as anxiety, depression, and reduced quality of life. Greater glycemic variability (GV) is associated with a higher risk of hypoglycemia and diabetes complications. Young adults are particularly at risk because they report greater FOH and have poorer glycemic control. A major gap exists in how to manage FOH as a crucial component of diabetes self-care. Our overall objective is to reduce FOH and improve diabetes self-management, glycemic control, and variability in young adults with T1DM. We specifically aim to: (1) Determine the feasibility of an 8-week CBT-based intervention to reduce FOH and (2) obtain means and standard deviations of group differences from baseline to program completion on the outcomes of FOH, self-management, glycemic control and glycemic variability in young adults with T1DM who experience FOH. To achieve these aims, we propose a randomized control pilot trial in 10 young adults aged 18 to 30 years with T1DM. Participants will be screened for FOH levels. Eligible subjects will be randomized to the intervention (Fear Reduction Efficacy Evaluation [FREE]) program or attention control group. A 1-week run-in phase is planned, with baseline measures of FOH and 24-hour real-time continuous glucose monitoring recordings (RT-CGM) to calculate GV for both groups. The intervention group will participate in eight weekly one-hour sessions using a cognitive behavioral therapy (CBT) and exposure treatment for specific fears. RT-CGM and a daily FOH diary will be used as feedback cues. The control group will wear a 24-hour RT-CGM device during the same 8-week period and return for weekly RT-CGM site changes by study staff. At completion, FOH will be measured, and RT-CGM recordings will be analyzed to determine within-group and between-group differences. The findings from this proposed study will serve as the foundation for a larger clinical trial to reduce FOH and improve self-management, glycemic control, and variability. Meeting these goals will have important clinical implications to reduce diabetes complications and improve quality of life in young adults with T1DM.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes ≥ 1 year
* receive medical care from an endocrinologist
* use insulin pump therapy
* have self-reported fear of hypoglycemia (FOH;screening questionnaire)

Exclusion Criteria:

* pregnant or breastfeeding
* actively treated for a mental health condition
* have a co-existing chronic illness or taking medications (excluding insulin) that may influence diabetes self-management or glycemic variability

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Martyn-Nemeth, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited through Chicago metropolitan area university medical centers, local diabetes websites, and organizations using flyers, e-announcements, and recruitment letters.
Period: Overall Study
Arm/Group | FREE Group | Control Group
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FREE Group | Control Group | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Hypoglycemia Fear Survey II - Worry subscale [Mean (Standard Deviation); unit: units on a scale] — Worry subscale of the Hypoglycemia Survey II was used to measure fear of hypoglycemia. This is an 18-item, 5-point [0-4] Likert scale that measures situation specific worries about hypoglycemia. The items are summed to provide an overall fear of hypoglycemia (worry) score. Scores may range from 0-72. Higher numbers indicate greater fear of hypoglycemia. The score is used as a continuous variable.
  units on a scale | 36.6 (18.4) | 38.8 (6.0) | 37.7 (12.9)
Diabetes Self-management Questionnaire [Mean (Standard Deviation); unit: units on a scale] — This is a 27-item, 4-point Likert scale questionnaire that measures diabetes self-management behavior. Scores may range from 0-81. The items are summed for an overall cotinuous scale score. Higher scores indicate better self-management behavior.
  units on a scale | 56.2 (13.2) | 52.2 (11.5) | 54.2 (11.9)
A1C [Mean (Standard Deviation); unit: percentage] — Hemoglobin A1c % represents the average blood glucose over a 3-month period. This variable was used as a continuous variable.
  percentage | 7.2 (1.29) | 7.96 (1.3) | 7.58 (1.28)
Glycemic variability [Mean (Standard Deviation); unit: mg/dL] | 66.04 (16.7) | 79.3 (12.9) | 71.03 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemia Fear Scale Score (HFS_2)
Description: A reliable and valid psychological scale. It is a 5-point Likert scale [0-4], that is summed for a single total continuous scale score. Scores may range from 0-72. Higher numbers indicate greater fear of hypoglycemia.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FREE Group | Control Group
Number analyzed (Participants) | 5 | 5
units on a scale | 21.4 (10.9) | 38.6 (8.2)

2. Secondary Outcome: Diabetes Self-Management Questionnaire Scale Score (DSMQ)
Description: A reliable and valid behavioral scale, provides total continuous scale score, ranging from 0-81, higher numbers indicate better self-management.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FREE Group | Control Group
Number analyzed (Participants) | 5 | 5
units on a scale | 58.7 (12.6) | 50.6 (12.1)

3. Secondary Outcome: Glycemic Control, the Average Blood Glucose Over a 2-3 Month Period of Time.
Description: Hemoglobin A1c represents the average blood glucose over a 2-3 month period and is an index of glycemic control. The American Diabetes Association recommends a hemoglobin A1C below 7% for most people with diabetes. Higher percentages indicate higher average blood glucose levels.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | FREE Group | Control Group
Number analyzed (Participants) | 5 | 5
percentage | 6.94 (1.29) | 7.66 (1.02)

4. Secondary Outcome: Glycemic Variability
Description: Twenty-four hour fluctuations in glucose measured by a continuous glucose monitor that provides interstitial glucose readings every 5 minutes. This is a continuous measure. A higher standard deviation reflects greater glycemic variability.
Time Frame: 8 weeks
Population: Same as above
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FREE Group | Control Group
Number analyzed (Participants) | 5 | 5
mg/dL | 73.0 (13.8) | 73.3 (11.8)

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | FREE Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT03165786/Prot_SAP_000.pdf